CLINICAL TRIAL: NCT03364244
Title: Revatio Special Investigation - Investigation for Long-Term Use of Revatio in Pediatric Patients
Brief Title: Revatio Special Investigation for Long-term Use in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Viatris Pharmaceuticals Japan Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: A1481319
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Revatio; Pulmonary arterial hypertension; Pediatric patients
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sildenafil: Pediatric patients receiving Revatio
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — [REVATIO® Tablets / REVATIO® OD Film] Adults Usually, sildenafil 20 mg is orally given three times daily. Children aged 1 year or older In children weighing 20 kg or more: Usually, sildenafil 20 mg is orally given three times daily.
  [REVATIO® Dry Syrup for Suspension] Adults Usually, sildenafil 20 mg is orally given three times daily. Children aged 1 year or older In children weighing 8 kg or more but less than 20 kg: Usually, sildenafil 10 mg is orally given three times daily.
  In children weighing 20 kg or more: Usually, sildenafil 20 mg is orally given three times daily.

SUMMARY:
Secondary data collection study: safety and effectiveness of Revatio in pediatric patients under Japanese medical practice

DETAILED DESCRIPTION:
The objective of this study is to obtain the information on dosage and administration, safety, and efficacy of Revatio when it is administered for a long period of time (1 year) under the actual use after the approval of the dosage and administration in pediatric patients (aged 1 year or older, weighed 8 kg or more) .

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0 to under 15 years who were confirmed to have received Revatio after the approval date of dosage and administration of Revatio for pediatric patients.

Exclusion Criteria:

* None.

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 0 to under 15 years who were confirmed to have received Revatio after the approval date of dosage and administration of Revatio for pediatric patients
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | 1 year (52 week) after observation start date
  The number of cases of adverse drug reactions during the observation period and their ratio are tabulated for each SOC and PT.
Effictiveness rate for physician's evaluation of this product | 1 year (52 week) after observation start date
  For the judgment of clinical effect at each evaluation time point (16th week, 52nd week and final evaluation time), the frequency (number of cases) and the ratio of each classification (valid, invalid, undecidable) are calculated.

SECONDARY OUTCOMES:
the dosage and administration under the actual use (including patients under the age of 1 year, weighing below 8 kg) | 1 year (52 week) after observation start date
  The mean doses at the initial , 16th, 52nd, and final evaluations are summarized for each newly treated case since dosage approval and continued case before dosage approval.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Nachankar, Study Director — Viatris Inc.
Locations (1):
- Viatris Pharmaceuticals Japan Inc., 5-11-2; Toranomon, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Sponsor will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A1481319